CLINICAL TRIAL: NCT05056246
Title: A Phase I, Open-label, Randomized, Parallel-arm, Single-dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of AMG 133 Administered Subcutaneously in Healthy Japanese and Caucasian Subjects
Brief Title: Study of AMG 133 Administered Subcutaneously in Healthy Japanese and Caucasian Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20200290
Record Dates: First submitted 2021-09-15; First posted 2021-09-24 (Actual); Results first posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-01

CONDITIONS: Healthy Participants
Keywords: Maridebart Cafraglutide; Japanese participants; Caucasian participants; AMG 133

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Japanese Participants: AMG 133 Low Dose (Experimental): Healthy Japanese participants will receive the low dose of AMG 133 as a SC injection on Day 1 of the study.
  Interventions: Drug: AMG 133
- Japanese Participants: AMG 133 Medium Dose (Experimental): Healthy Japanese participants will receive the medium dose of AMG 133 as a SC injection on Day 1 of the study.
  Interventions: Drug: AMG 133
- Japanese Participants: AMG 133 High Dose (Experimental): Healthy Japanese participants will receive the high dose of AMG 133 as a SC injection on Day 1 of the study.
  Interventions: Drug: AMG 133
- Caucasian Participants: AMG 133 Medium Dose (Experimental): Healthy Caucasian participants will receive the medium dose of AMG 133 as a SC injection on Day 1 of the study.
  Interventions: Drug: AMG 133
- Caucasian Participants: AMG 133 High Dose (Experimental): Healthy Caucasian participants will receive the high dose of AMG 133 as a SC injection on Day 1 of the study.
  Interventions: Drug: AMG 133

INTERVENTIONS:
Drug: AMG 133 — Solution for SC injection
  Other Names: maridebart cafraglutide

SUMMARY:
The primary objective of this study is to evaluate the pharmacokinetics (PK) of AMG 133 after single subcutaneous (SC) administration in healthy Japanese and Caucasian participants.

ELIGIBILITY:
Key Inclusion Criteria:

1. Healthy male or female participants between 18 and 65 years of age (inclusive) at the time of Screening (Japanese participants must be first-generation Japanese)
2. In good health, determined by no clinically significant findings from medical history, physical examination, ECG, vital signs measurements, and clinical laboratory evaluations
3. Body mass index between 18 and 30 kg/m^2 at the time of Screening
4. Females of nonchildbearing potential

Key Exclusion Criteria:

1. History or evidence, at Screening or Check-in, of clinically significant disorder, condition, or disease
2. History or current signs or symptoms of cardiovascular disease
3. History or evidence of clinically significant arrhythmia at Screening, including any clinically significant findings on the ECG taken at Check-in
4. History of hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance
5. Positive hepatitis B or hepatitis C panel and/or positive human immunodeficiency virus test at Screening
6. History of alcoholism or drug/chemical abuse within 1 year prior to Check-in
7. Use of tobacco- or nicotine-containing products within 6 months prior to Check-in
8. Positive test for illicit drugs, cotinine (tobacco or nicotine use), and/or alcohol use at Screening or Check-in
9. Female participants with a positive pregnancy test at Screening or Check-in
10. Female participants lactating/breastfeeding or who plans to breastfeed during the study through 90 days after the end of study (EOS) visit
11. Donation of blood from 3 months prior to Check-in, plasma from 2 weeks prior to Check-in, or platelets from 6 weeks prior to Check-in
12. Unwilling to abide with study restrictions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2022-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- WCCT Global LLC, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy Japanese and Caucasian participants were enrolled at a single center in the United States between 10 September 2021 and 08 April 2022.
Pre-assignment Details: A total of 34 participants were enrolled and randomized in the study. All 34 participants were dosed in accordance with the protocol.
Groups:
- Japanese Participants: AMG 133 Low Dose: Healthy Japanese participants received the low dose of AMG 133 as a subcutaneous (SC) injection on Day 1 of the study.
- Japanese Participants: AMG 133 Medium Dose: Healthy Japanese participants received the medium dose of AMG 133 as a SC injection on Day 1 of the study.
- Japanese Participants: AMG 133 High Dose: Healthy Japanese participants received the high dose of AMG 133 as a SC injection on Day 1 of the study.
- Caucasian Participants: AMG 133 Medium Dose: Healthy Caucasian participants received the medium dose of AMG 133 as a SC injection on Day 1 of the study.
- Caucasian Participants: AMG 133 High Dose: Healthy Caucasian participants received the high dose of AMG 133 as a SC injection on Day 1 of the study.
Period: Overall Study
Arm/Group | Japanese Participants: AMG 133 Low Dose | Japanese Participants: AMG 133 Medium Dose | Japanese Participants: AMG 133 High Dose | Caucasian Participants: AMG 133 Medium Dose | Caucasian Participants: AMG 133 High Dose
Started | 6 | 7 | 7 | 7 | 7
Received AMG 133 | 6 | 7 | 7 | 7 | 7
Completed | 6 | 6 | 7 | 5 | 6
Not Completed | 0 | 1 | 0 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: Included all participants who received at least 1 dose of AMG 133.
Groups:
- Japanese Participants: AMG 133 Low Dose: Healthy Japanese participants received the low dose of AMG 133 as a SC injection on Day 1 of the study.
- Total: Total of all reporting groups
Arm/Group | Japanese Participants: AMG 133 Low Dose | Japanese Participants: AMG 133 Medium Dose | Japanese Participants: AMG 133 High Dose | Caucasian Participants: AMG 133 Medium Dose | Caucasian Participants: AMG 133 High Dose | Total
Number analyzed (Participants) | 6 | 7 | 7 | 7 | 7 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (4.80) | 55.0 (5.35) | 52.9 (13.90) | 43.0 (14.59) | 49.0 (11.93) | 51.3 (11.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 4 | 1 | 2 | 13
  Male | 3 | 4 | 3 | 6 | 5 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 2 | 4 | 6
  Not Hispanic or Latino | 6 | 7 | 7 | 5 | 3 | 28
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 0 | 0 | 0 | 7 | 7 | 14
  Japanese | 6 | 7 | 7 | 0 | 0 | 20

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Intact AMG 133
Description: Blood samples were collected at specific times during the study for the measurement of plasma concentrations of intact and total AMG 133 by a laboratory.
Time Frame: Day 1 pre-dose and 24, 48, 72, 96, 120, 144, 168, 336, 504, 672, 1008, 1344, 1680, 2184, and 2856 hours post-dose
Population: Pharmacokinetic (PK) Population: Included all participants who received at least 1 dose of AMG 133 and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Japanese Participants: AMG 133 Low Dose | Japanese Participants: AMG 133 Medium Dose | Japanese Participants: AMG 133 High Dose | Caucasian Participants: AMG 133 Medium Dose | Caucasian Participants: AMG 133 High Dose
Number analyzed (Participants) | 6 | 7 | 7 | 7 | 6
μg/mL | 12.3 (57.3) | 22.7 (24.1) | 44.9 (34.6) | 22.5 (33.9) | 55.0 (26.7)

2. Primary Outcome: Cmax of Total AMG 133
Description: as for outcome 1
Time Frame: Day 1 pre-dose and 24, 48, 72, 96, 120, 144, 168, 336, 504, 672, 1008, 1344, 1680, 2184, and 2856 hours post-dose
Population: PK Population: Included all participants who received at least 1 dose of AMG 133 and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Japanese Participants: AMG 133 Low Dose | Japanese Participants: AMG 133 Medium Dose | Japanese Participants: AMG 133 High Dose | Caucasian Participants: AMG 133 Medium Dose | Caucasian Participants: AMG 133 High Dose
Number analyzed (Participants) | 6 | 7 | 7 | 7 | 6
μg/mL | 13.2 (56.3) | 24.8 (25.6) | 48.4 (32.0) | 20.8 (24.5) | 58.7 (24.8)

3. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Time of Last Quantifiable Concentration (AUClast) of Intact AMG 133
Description: as for outcome 1
Time Frame: Day 1 pre-dose and 24, 48, 72, 96, 120, 144, 168, 336, 504, 672, 1008, 1344, 1680, 2184, and 2856 hours post-dose
Population: PK Population: Included all participants who received at least 1 dose of AMG 133 and had evaluable PK data. Only participants with available data are included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Japanese Participants: AMG 133 Low Dose | Japanese Participants: AMG 133 Medium Dose | Japanese Participants: AMG 133 High Dose | Caucasian Participants: AMG 133 Medium Dose | Caucasian Participants: AMG 133 High Dose
Number analyzed (Participants) | 6 | 6 | 7 | 5 | 6
h*ug/mL | 10600 (45.2) | 19400 (36.0) | 33500 (20.5) | 17200 (42.4) | 35700 (31.1)

4. Primary Outcome: AUClast of Total AMG 133
Description: as for outcome 1
Time Frame: Day 1 pre-dose and 24, 48, 72, 96, 120, 144, 168, 336, 504, 672, 1008, 1344, 1680, 2184, and 2856 hours post-dose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Japanese Participants: AMG 133 Low Dose | Japanese Participants: AMG 133 Medium Dose | Japanese Participants: AMG 133 High Dose | Caucasian Participants: AMG 133 Medium Dose | Caucasian Participants: AMG 133 High Dose
Number analyzed (Participants) | 6 | 6 | 7 | 5 | 6
h*ug/mL | 14800 (41.8) | 28300 (37.2) | 47700 (21.1) | 20800 (41.4) | 49600 (30.9)

5. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinity (AUCinf) of Intact AMG 133
Description: as for outcome 1
Time Frame: Day 1 pre-dose and 24, 48, 72, 96, 120, 144, 168, 336, 504, 672, 1008, 1344, 1680, 2184, and 2856 hours post-dose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Japanese Participants: AMG 133 Low Dose | Japanese Participants: AMG 133 Medium Dose | Japanese Participants: AMG 133 High Dose | Caucasian Participants: AMG 133 Medium Dose | Caucasian Participants: AMG 133 High Dose
Number analyzed (Participants) | 6 | 6 | 7 | 5 | 6
h*ug/mL | 10700 (44.9) | 19600 (36.4) | 33900 (20.4) | 17300 (43.3) | 36000 (31.6)

6. Primary Outcome: AUCinf of Total AMG 133
Description: as for outcome 1
Time Frame: Day 1 pre-dose and 24, 48, 72, 96, 120, 144, 168, 336, 504, 672, 1008, 1344, 1680, 2184, and 2856 hours post-dose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Japanese Participants: AMG 133 Low Dose | Japanese Participants: AMG 133 Medium Dose | Japanese Participants: AMG 133 High Dose | Caucasian Participants: AMG 133 Medium Dose | Caucasian Participants: AMG 133 High Dose
Number analyzed (Participants) | 6 | 6 | 7 | 5 | 6
h*ug/mL | 15600 (40.5) | 30100 (39.2) | 50100 (21.8) | 21800 (45.4) | 51500 (32.5)

7. Secondary Outcome: Number of Participants Who Experienced a Treatment-emergent Adverse Event (TEAE)
Description: A TEAE was defined as any untoward medical occurrence in a clinical study participant irrespective of a causal relationship with AMG 133 that started during or after dosing, or started prior to dosing and increased in severity after dosing.
  Clinically significant changes from baseline in clinical laboratory tests, 12-lead electrocardiograms (ECGs) and vital signs were also reported as TEAEs.
Time Frame: Day 1 to Day 120
Population: Safety Population: Included all participants who received at least 1 dose of AMG 133.
Measure: Count of Participants; unit: Participants
Arm/Group | Japanese Participants: AMG 133 Low Dose | Japanese Participants: AMG 133 Medium Dose | Japanese Participants: AMG 133 High Dose | Caucasian Participants: AMG 133 Medium Dose | Caucasian Participants: AMG 133 High Dose
Number analyzed (Participants) | 6 | 7 | 7 | 7 | 7
Participants | 6 | 6 | 7 | 7 | 7

8. Secondary Outcome: Number of Participants With a Positive Anti-AMG 133 Binding Antibody Result
Description: Blood samples were collected at specific times during the study for the measurement of anti-AMG 133 binding antibodies from participants who received AMG 133.
Time Frame: Days 1, 15, 29, 57 and 120
Population: Safety Population: Included all participants who received at least 1 dose of AMG 133.
Measure: Count of Participants; unit: Participants
Arm/Group | Japanese Participants: AMG 133 Low Dose | Japanese Participants: AMG 133 Medium Dose | Japanese Participants: AMG 133 High Dose | Caucasian Participants: AMG 133 Medium Dose | Caucasian Participants: AMG 133 High Dose
Number analyzed (Participants) | 6 | 7 | 7 | 7 | 7
Participants | 3 | 3 | 3 | 1 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality was collected from enrolment to end of study (median [min,max]: 4.42 months [1.51, 5.42 months]. Serious adverse events and other adverse events were collected from Day 1 to Day 120.
Arm/Group | Japanese Participants: AMG 133 Low Dose | Japanese Participants: AMG 133 Medium Dose | Japanese Participants: AMG 133 High Dose | Caucasian Participants: AMG 133 Medium Dose | Caucasian Participants: AMG 133 High Dose
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7 | 0/7 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7 | 1/7 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 6/6 | 6/7 | 7/7 | 7/7 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Japanese Participants: AMG 133 Low Dose (N=6) | Japanese Participants: AMG 133 Medium Dose (N=7) | Japanese Participants: AMG 133 High Dose (N=7) | Caucasian Participants: AMG 133 Medium Dose (N=7) | Caucasian Participants: AMG 133 High Dose (N=7)
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Japanese Participants: AMG 133 Low Dose (N=6) | Japanese Participants: AMG 133 Medium Dose (N=7) | Japanese Participants: AMG 133 High Dose (N=7) | Caucasian Participants: AMG 133 Medium Dose (N=7) | Caucasian Participants: AMG 133 High Dose (N=7)
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Bowel movement irregularity (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 5 | 6 | 7 | 7 | 7
Vomiting (Gastrointestinal disorders) | 4 | 6 | 7 | 7 | 7
Chills (General disorders) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 2 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 1
Acarodermatitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Asymptomatic COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 2 | 2
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Pancreatic enzymes increased (Investigations) | 0 | 0 | 0 | 1 | 1
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1 | 1 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 3 | 5 | 3 | 3
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 3
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2021-08-24): https://cdn.clinicaltrials.gov/large-docs/46/NCT05056246/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-18): https://cdn.clinicaltrials.gov/large-docs/46/NCT05056246/SAP_001.pdf